CLINICAL TRIAL: NCT04441099
Title: A First-in-Human, Phase 1/2 Study of NBE-002, an Anti-ROR1 Antibody Drug Conjugate, in Patients With Advanced Solid Tumors
Brief Title: NBE-002 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: End of Program
Sponsor: NBE-Therapeutics AG (Industry)
Collaborators: Cmed Clinical Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NBE-002-01
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor; Advanced Cancer; Triple Negative Breast Cancer
Keywords: ROR1; Antibody-drug Conjugate; Carcinoma; Cancer; Solid Tumor; Sarcoma; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma; Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-escalation Cohort (DEC) (Experimental): Escalating doses of NBE-002 depending on cohort at enrollment.
  Interventions: Drug: NBE-002
- Safety-expansion Cohort (SEC) (Experimental): Dose to be determined based on DEC.
  Interventions: Drug: NBE-002
- Expansion Cohort 1 (EC1) (Experimental): Dose to be determined based on DEC and SEC.
  Interventions: Drug: NBE-002
- Expansion Cohort 2 (EC2) (Experimental): Dose to be determined based on DEC and SEC.
  Interventions: Drug: NBE-002

INTERVENTIONS:
Drug: NBE-002 — NBE-002 will be given intravenously on Day 1 of repeated 28-day cycles.

SUMMARY:
This first-in-human study will evaluate the recommended dose for further clinical development, safety, tolerability, anti-tumor activity, immunogenicity, pharmacokinetics and pharmacodynamics of NBE-002, a novel anti-ROR1 antibody-drug conjugate, in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Phase 1, DEC and SEC: patients with histologically or cytologically confirmed advanced solid tumor (carcinoma or sarcoma), who have progressive disease, have undergone systemic therapy for advanced disease, and for whom no standard therapy is available
* Phase 2, EC1: patients with histologically or cytologically confirmed advanced triple-negative breast cancer, who have progressive disease, and have undergone no more than three prior lines of systemic therapy for advanced disease
* Phase 2, EC2: patients with histologically or cytologically confirmed advanced solid tumor (carcinoma or sarcoma) other than TNBC, who have progressive disease, and have undergone no more than three prior lines of systemic therapy for advanced disease
* Availability of pretreatment tumor tissue
* Phase 1, DEC and SEC: at least one measurable or non-measurable lesion as per RECIST v1.1
* Phase 2, EC1 and EC2: at least one measurable lesion as per RECIST v1.1
* Phase 1, DEC and SEC: Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Phase 2, EC1 and EC2: ECOG performance status of 0 or 1
* Adequate function of bone marrow, liver, kidneys, heart; adequate coagulation profile
* Both male and female patients must agree to use effective contraceptive methods
* Women of child-bearing potential (WCBP) must have a negative serum pregnancy test
* Patients must be willing and able to sign the informed consent form, and to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Prior treatment with any agent targeting ROR1
* Presence of active central nervous system (CNS) metastasis
* Persistent toxicities from previous systemic anti-neoplastic treatments of Grade > 1 (or Grade > 2 for neurotoxicity)
* Systemic anti-neoplastic therapy within five half-lives or four weeks (six weeks for nitrosourea and mitomycin-C), whichever is shorter, prior to first dose of the study drug
* Wide-field radiotherapy within four weeks, or focal radiation for analgesic purpose or for lytic lesions at risk of fracture within two weeks prior to first dose of the study drug, or no recovery from side effects of such intervention
* Major surgery within four weeks prior to first dose of the study drug, or no recovery from side effects of such intervention
* Prior allogeneic bone marrow transplantation
* Significant cardiac disease
* History of thromboembolic or cerebrovascular events within six months prior to first dose of the study drug
* Acute and/or clinically significant bacterial, fungal or viral infection
* Concomitant use of systemic steroids at dose of >10 mg of prednisone or its equivalent per day
* Concurrent participation in another investigational clinical trial
* Pregnant or breast-feeding females
* Other conditions that prevent the patient from giving informed consent or participating in the trial, or that may increase the risk associated with the study participation, or that may interfere with the interpretation of the study results
* Prior history of malignancy other than inclusion diagnosis within three years prior to first dose of the study drug
* Prior treatment with cumulative lifetime dose of anthracycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) (Phase 1) | Up to 48 months
  The RP2D will be determined using dose limiting toxicities (DLTs) and all other available study data
Anti-tumor Activity (Phase 2) | Up to 60 months
  Anti-tumor activity will be assessed by Response Evaluation Criteria in Solid Tumours (RECIST) v1.1

SECONDARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | Up to 60 months
  Safety and tolerability profile will be assessed by Common Terminology Criteria for Adverse Events v5.0 and summarized by type, frequency, and severity of adverse events
Preliminary Anti-tumor Activity (Phase 1) | Up to 48 months
  Preliminary anti-tumor activity will be assessed by Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
Concentrations of NBE-002 | Up to 60 months
  Pharmacokinetic profile will be characterized by concentrations of NBE-002
Concentrations of NBE-002-reactive antibodies | Up to 60 months
  Immunogenicity profile will be characterized by concentrations of NBE-002-reactive antibodies

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sarah Cannon Research Institute - TN Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No